CLINICAL TRIAL: NCT04259086
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of DaxibotulinumtoxinA for Injection (DAXI for Injection) for the Combined Treatment of Upper Facial Lines (Glabellar Lines, Dynamic Forehead Lines and Lateral Canthal Lines)
Brief Title: Efficacy and Safety of DaxibotulinumtoxinA (DAXI) for Injection for Treatment of Upper Facial Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1920201
Record Dates: First submitted 2019-12-19; First posted 2020-02-06 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Upper Facial Lines (Glabellar Lines, Forehead Lines, & Lateral Canthal Lines)
Keywords: Lateral Canthal Wrinkle; crow's feet lines; LCL; Forehead Lines; Glabellar Lines; Frown Lines; Upper facial lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DAXI 40 U GL / 32 U FHL / 48 U LCL (Experimental): DaxibotulinumtoxinA for injection for the treatment of moderate to severe Glabellar Lines (GL), Forehead Lines (FHL), & Lateral Canthal Lines (LCL)
  Interventions: Drug: DaxibotulinumtoxinA for injection

INTERVENTIONS:
Drug: DaxibotulinumtoxinA for injection — Intramuscular injection

SUMMARY:
This is a Phase 2, multicenter, open-label, single-arm study to evaluate the efficacy and safety of DaxibotulinumtoxinA for injection (DAXI for injection) in the treatment of Glabellar Lines (GL), Dynamic Forehead Lines (FHL), and Lateral Canthal Lines(LCL)

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines and local laws, including authorization to release health information, signed prior to any study procedures being performed
2. Be outpatient, male or female subjects, in good general health, 18 years of age or older
3. Have a score of moderate (2) or severe (3) Glabellar Lines during maximum contraction as assessed by the Investigator Global Assessment-Frown Wrinkle Severity (IGA-FWS) and Patient Frown Wrinkle Severity (PFWS)
4. Have a score of moderate (2) or severe (3) Forehead Lines during maximum contraction as assessed by the Investigator Global Assessment Forehead Wrinkle Severity (IGA-FHWS) and Patient Forehead Wrinkle Severity (PFHWS)
5. Have a score of moderate (2) or severe (3) Lateral Canthal Lines at maximum contraction as assessed by the Investigator Global Assessment of Lateral Canthal Wrinkle Severity (IGA-LCWS) and Patient Lateral Canthal Wrinkle Severity (PLCWS) (scores must be consistent bilaterally for each scale considered separately)
6. Able to understand the requirements of the study and be willing and able to follow all study procedures, attend all scheduled visits, comprehend and complete the questionnaires without outside assistance and successfully complete the study

Exclusion Criteria:

1. Active skin disease, infections, or inflammation at the injection sites
2. Planned or anticipated need for surgery or hospitalization through the end of the study
3. Pregnant, nursing, or planning a pregnancy during the study; or is a Women of Child Bearing Potential (WOCBP) but is not willing to use an effective method of contraception
4. Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Site 1, Manhattan Beach, California
  - Site 3, San Diego, California
  - Site 7, Santa Monica, California
  - Site 5, Coral Gables, Florida
  - Site 2, Chestnut Hill, Massachusetts
  - Site 6, New York, New York
- Canada (2):
  - Site 4, Vancouver, British Columbia
  - Site 8, Toronto, Ontario

REFERENCES:
- [Derived] Dover JS, Humphrey SD, Lorenc ZP, Shamban A, Gross TM, Rubio RG, Vitarella D. Treatment of Upper Facial Lines With DaxibotulinumtoxinA for Injection: Results From an Open-Label Phase 2 Study. Dermatol Surg. 2023 Jan 1;49(1):60-65. doi: 10.1097/DSS.0000000000003637. Epub 2022 Nov 28. PMID 36533798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DAXI 40 U GL / 32 U FHL / 48 U LCL
Started | 48
Completed | 45
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | DAXI 40 U GL / 32 U FHL / 48 U LCL
Number analyzed (Participants) | 48
Age, Continuous [Mean (Full Range); unit: years] | 48.9 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 44
  Race: Black/African American | 3
  Race: Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With None or Mild in GL Severity at Maximum Frown
Description: The percentage of subjects achieving a score of 0 (none) or 1 (mild) in GL severity at maximum contraction (maximum frown) at Week 4 as assessed by the IGA-FWS
Time Frame: Week 4
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | DAXI 40 U GL / 32 U FHL / 48 U LCL
Number analyzed (Participants) | 48
Participants | 46

2. Primary Outcome: Percentage of Participants With None or Mild in FHL Severity at Maximum Eyebrow Elevation
Description: The percentage of subjects achieving a score of 0 (none) or 1 (mild) in FHL severity at maximum contraction (maximum eyebrow elevation) at Week 4 as assessed by the IGA-FHWS
Time Frame: Week 4
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | DAXI 40 U GL / 32 U FHL / 48 U LCL
Number analyzed (Participants) | 48
Participants | 46

3. Primary Outcome: Percentage of Participants With None or Mild in LCL Severity at Maximum Smile Effort
Description: The percentage of subjects achieving a score of 0 (none) or 1 (mild) in LCL severity at maximum contraction (maximum smile effort) at Week 4 as assessed by the IGA-LCWS
Time Frame: Week 4
Population: Evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | DAXI 40 U GL / 32 U FHL / 48 U LCL
Number analyzed (Participants) | 48
Participants | 44

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the entire study, up to 36 weeks after treatment.
Description: The safety population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs.
Arm/Group | DAXI 40 U GL / 32 U FHL / 48 U LCL
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 40 U GL / 32 U FHL / 48 U LCL (N=48)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 40 U GL / 32 U FHL / 48 U LCL (N=48)
Injection site erythema (General disorders) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (2):
  • Study Protocol (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT04259086/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04259086/SAP_001.pdf